CLINICAL TRIAL: NCT00166179
Title: Magnetic Resonance Imaging (MRI) Viability: Comparison of Myocardial Viability by Positron Emission Tomography and MRI
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Randolph E Patterson, Professor, Emory University
Other Study IDs: IRB00000292; 6-56550 (Other: Other)
Record Dates: First submitted 2005-09-13; First posted 2005-09-14 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Coronary Artery Disease
Keywords: CAD
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare cardiac MRI with positron emission tomography (PET) with fluorodeoxyglucose (FDG) to determine if cardiac MRI images are as good as, or better, than PET with FDG.

ELIGIBILITY:
Inclusion Criteria:

* PET-FDG ordered to assess myocardial viability

Exclusion Criteria:

* Contraindicated for MRI
* Pregnant
* Age <25 yrs

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age > 25 yrs, mean + SD = 60.3 + 10.2, 83% male, are patients referred by cardiologist or cardiac surgeon for assessment of myocardial viability by PET FDG.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2003-11; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Magnetic Resonance Imaging (MRI) Viability: Comparison of Myocardial Viability by Positron Emission Tomography and MRI | time of initial scans

SECONDARY OUTCOMES:
Compare size of regions of viable and non viable myocardium as % left ventricle by MRI vs. PET | at time of initial scans

CONTACTS AND LOCATIONS:
Overall Officials: Randolph Patterson, MD, Principal Investigator — Staff
Locations (1):
- Crawford Long Hospital, Atlanta, Georgia, United States